CLINICAL TRIAL: NCT02403245
Title: The Impact of a Social Stimulation on Social Interactions in Institutionalized People With Dementia
Brief Title: Social Interactions Between People With Dementia in Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paris West University Nanterre La Défense (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Jean-Bernard Mabire, psychologist and PhD psychologist Student, Paris West University Nanterre La Défense
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SID010
Record Dates: First submitted 2015-03-16; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Dementia; Social Interactions
Keywords: Social interactions; Dementia; Social stimulation; Direct observation
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychosocial stimulation (Experimental): One session of a social stimulation
  Interventions: Other: Psychosocial stimulation
- Control group (No Intervention): Residents are in a social controlled condition but without direct stimulation.

INTERVENTIONS:
Other: Psychosocial stimulation — Intervention consists in a session of social stimulation during about 40 minutes through where the speaker introduced himself to the residents and introduces the residents to each others. The date of the day was done to residents. Social stimulation consists here to an exercise about the four seasons. Residents are asked to mention the 4 seasons and to give all the characteristics they can about each season. Two exercises were proposed: 4 pictures of landscapes and residents were asked to tell which season is represent on the pictures and pictures of some fruits and residents tried to tell in which season we find the fruits. Finally, the psychologist speaks about the "four season" of the compositor Vivaldi and propose to the residents to listen some extracts of each pieces of music.
  Arms: Psychosocial stimulation

SUMMARY:
The aim of this study is to evaluate the direct impact of one session of social stimulation on social interactions of people with moderate dementia living in nursing home in comparison of one session without direct social stimulation.

DETAILED DESCRIPTION:
60 people with moderate dementia living in a french nursing homme participated in this study. Residents gave oral consent twice to participate. They were classified in groups of six residents taking into account socio-demographic and medical characteristics. Two experimental conditions were proposed : 1. a social stimulation session (36 residents) and 2. a control group without direct social stimulation (24 residents). Collected socio-demographic and medical characteristics are age, gender, timf of institutionalization, sociocultural level, marital status and diagnostic hypothesis. Before the study, scales and questionnaires were used to assess cognitive status with the Mini Mental State Examination (Folstein et al, 1975); functional abilities with Instrumental Activities of Daily Living (Lawton and Brody, 1969); depression with the Cornell Scale for Depression in Dementia (Alexopoulos et al, 1988); psychological and behavioural disorders with the Neuropsychiatric Inventory (Cummings et al, 1994); and the quality of life with the Alzheimer's Disease Related Quality of Life (Rabins et al, 1999).

Social interactions are video taped and analyzed in a grid of observation.

The aim of the study is to see if there is an impact on social interactions after just one social stimulation session compared to a control group situation. Expected results are that residents of the social stimulation group will have more social interactions between us than the resident of the control group.

ELIGIBILITY:
Inclusion Criteria:

* presence of a diagnostic of dementia in medical report and a MMSE score between 9 and 20.

Exclusion Criteria:

* arrival in the institution dating less than six months
* invalidating visual or hearing disorders
* phasic disorders not allowing a minimum of communication
* significant behavioural disorders (which can disturb the meeting)
* residents not fluent in French language

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Observed social behaviours | during 8 minutes before the session a
  social behaviours of residents observed and listed in an observations grid to analyze the results from observation in terms of components of behaviours expressed in means of observed behaviours.
Observed social behaviours | during 8 minutes after the session
  social behaviours of residents observed and listed in an observations grid to analyze the results from observation in terms of components of behaviours expressed in means of observed behaviours.

SECONDARY OUTCOMES:
Cognitive Status | Baseline
  Scale of the Mini Mental State of examination scored on 30 points.
Functional abilities | Baseline
  Scale of the Instrumental Activities of Daily Living scored on 14 points. More the score is high more the people is independent in daily living.
Depression | Baseline
  Cornell Scale for Depression in Dementia scored on 38 points. More the score os high more the people is depressed with a threshold score of 10.
Psychological and behaviors disorders | Baseline
  Neuropsychiatric Inventory : hetero-evaluation of the psychological and behavioural disorders in 12 domains with the frequency of occurrence of the disorder, the intensity and the resounding on caregivers.
Quality of life | Baseline
  Hetero-evaluation scale named Alzheimer's Disease Related Quality of life expressed in percentage. A high score means a good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard Mabire, Principal Investigator — University Paris Ouest - EA 4430 - 200, Avenue de la République - 92001 Nanterre cedex